CLINICAL TRIAL: NCT00418691
Title: Assessing the Efficacy of Immediate Release Methylphenidate, Sustained Release Methylphenidate and Modafinil for Patients With Brain Tumors
Brief Title: Effects of Methylphenidate Versus Sustained Release Methylphenidate on Cognitive Functioning
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Closed early due to slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0925
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Brain Tumor
Keywords: Brain Tumor; Methylphenidate; Ritalin; Modafinil; Provigil; Fatigue; Concentration
MeSH Terms: conditions — Brain Neoplasms; Fatigue | interventions — Methylphenidate; Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Immediate Release (IR) Methylphenidate (Active Comparator): 10 mg by mouth (PO) twice daily for 4 Weeks
  Interventions: Drug: IR Methylphenidate
- Sustained Release (SR) Methylphenidate (Active Comparator): 200 mg PO once daily for 4 Weeks
  Interventions: Drug: SR Methylphenidate
- Modafinil (Active Comparator): 18 mg PO once daily for 4 Weeks
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: IR Methylphenidate — 10 mg by mouth (PO) twice daily x 4 Weeks
  Other Names: Ritalin
  Arms: Immediate Release (IR) Methylphenidate
Drug: Modafinil — 200 mg PO Once Daily x 4 Weeks
  Other Names: Provigil
  Arms: Modafinil
Drug: SR Methylphenidate — 18 mg PO Once Daily x 4 Weeks
  Other Names: Ritalin
  Arms: Sustained Release (SR) Methylphenidate

SUMMARY:
Primary Objective:

* To assess the efficacy of immediate release methylphenidate, sustained release methylphenidate, and the novel vigilance enhancing drug modafinil for the improvement of cognitive functioning in patients with brain tumors.

DETAILED DESCRIPTION:
All three drugs used in this clinical research study are widely used stimulants to help cancer patients who have fatigue and problems with concentration.

Before treatment starts, you will have a physical exam, including measurement of blood pressure, and neuropsychological and symptom evaluations. The neuropsychological evaluation is made up of tests of attention, memory, speech, and other brain functions, and takes about 30 minutes to complete. The other test evaluates symptoms you may be experiencing, such as fatigue or depression, and takes about 10 minutes to complete.

You will be randomly assigned (as in the toss of a coin) to one of three treatment groups. Participants in the first group will receive Immediate Release (IR) methylphenidate. Participants in the second group will receive Sustained Release (SR) methylphenidate. Participants in the third group will receive modafinil. There is an equal chance of being assigned to any of the groups. After you are randomized, you will contact the M. D. Anderson pharmacy to receive your assigned medication. You will receive a total of 5 weeks worth of medication. The extra week of medication is to allow for buffer should there be any conflict in rescheduling the follow-up evaluation.

IR methylphenidate is a pill taken twice a day. Both SR methylphenidate and modafinil are pills taken once a day. The amount of the medicine is the same for all three groups. You will take the medication every day for a total of 4 weeks.

You will be asked to complete a study calendar, which will be provided by the research staff. In the study calendar, you will be asked to initial after you take the study drug each day, and to record any side effects you may experience. You will be required to return the completed study calendar at the final evaluation visit, along with the empty bottles and any of the study drugs that may be left over.

You will remain on treatment for 4 weeks and return for a final evaluation. A follow-up neuropsychological evaluation and evaluation of symptoms will be performed. At the end of the study treatment period, you will be allowed to remain on active treatment if you wish to. You can discuss with your doctor whether to continue on the same medication or to try another one.

This is an investigational study. All of the study drugs are FDA approved and currently are used to help brain tumor patients. A total of 75 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with a brain tumor, either primary or metastatic
2. Patient had prior radiation treatment to the brain
3. Patient is > or = 18 years of age
4. Patient has a Karnofsky performance status (KPS) performance of 70 at baseline
5. Patient is using acceptable birth control methods. Female participants (if of child bearing age and sexually active) and male participants (if sexually active with a partner of child-bearing potential) must use medically acceptable methods of birth control, including abstinence, birth control pills, diaphragm with spermicide, condom with foam or spermicide, vaginal spermicidal suppository or surgical sterilization.
6. Patient must speak and understand English or Spanish
7. Patient has reported cognitive decline and is being considered for stimulant therapy by their neurologist
8. Patient has provided written informed consent to participate in the study prior to enrollment to the study

Exclusion Criteria:

1. History of hypersensitivity reaction to methylphenidate or modafinil
2. History of severe headaches, glaucoma, major psychiatric diagnosis, narcolepsy, Tourette's syndrome, marked anxiety, tension or agitation
3. History of clinically significant pulmonary or cardiac disease
4. Uncontrolled hypertension: has not been on a stable treatment dose for the past month, or has a systolic pressure consistently greater than 140 mm Hg or diastolic pressure consistently greater than 90 mm Hg
5. Patients with uncontrolled seizures will be excluded
6. Current use of illicit drugs or history of alcohol or drug abuse and/or abuse potential
7. Moderate to severe depression (> 20 on Beck Depression Inventory II)
8. If taking antidepressants, patient must be on a stable dose
9. Currently taking psychostimulants, Monoamine oxidase (MAO) inhibitors, or anticoagulants
10. Current use of the following herbals or supplements for fatigue relief (dehydroepiandrosterone (DHEA), S-Adenosyl methionine (SAME), ginkgo, ginseng, St. John's Wort)
11. Any coexisting medical condition or are taking any concomitant medication that is likely to interfere with the safe administration of methylphenidate. Any potential interactions or coexisting medical condition not specified by the protocol will be determined by the prescribing physician as being exclusionary or not.
12. Patients currently taking any erythropoietin type drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Wefel, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 2004 - April 2009. All recruiting done at UT MD Anderson Cancer Center, Neuro-Oncology Clinic.
Pre-assignment Details: Of the 34 registered patients, one enrolled patient did not join study and therefore was never included in any group assignment.
Groups:
- IR Methylphenidate: Immediate Release (IR) Methylphenidate 10 mg by mouth (PO) twice daily for 4 weeks
- SR Methylphenidate: Sustained Release (SR) Methylphenidate 200 mg PO once daily for 4 weeks
Period: Overall Study
Arm/Group | IR Methylphenidate | SR Methylphenidate | Modafinil
Started | 11 | 12 | 10
Completed | 9 | 10 | 5
Not Completed | 2 | 2 | 5
Not completed — Lost to Follow-up | 1 | 2 | 3
Not completed — Started new medication voiding entry | 0 | 0 | 1
Not completed — Progressive Disease | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IR Methylphenidate | SR Methylphenidate | Modafinil | Total
Number analyzed (Participants) | 11 | 12 | 10 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 7 | 30
  >=65 years | 0 | 0 | 3 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (10.0) | 41.2 (10.5) | 53.8 (12.9) | 46.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 4 | 16
  Male | 5 | 6 | 6 | 17
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 10 | 33

OUTCOME MEASURES:

1. Primary Outcome: Mean Processing Speed Change From Baseline in the Trail-making Test Part A Score
Description: 'Trail Making Test Part A' is a neuropsychological test of visual attention and task switching, administered to measure processing speed, timed as participants follow "trail" made by consecutive numbers (1,2,3, etc.). The test is finished as quickly as possible, and the time taken to complete the test used as the primary performance metric (in seconds). Maximum time allowed is 300 seconds. A lower change score indicates improvement. Participants tested before starting study medication and 4-5 weeks later while on study medication, reflected in a z score (deviations from population mean).
Time Frame: Baseline to 4-5 weeks on study medication
Population: Analysis were per protocol. The z-score reflects how many standard deviations above or below the population mean a raw score is for each participant.
Measure: Mean (Standard Deviation); unit: z-scores
Arm/Group | IR Methylphenidate | SR Methylphenidate | Modafinil
Number analyzed (Participants) | 11 | 12 | 10
z-scores | -4.7 (9.2) | 0.24 (1.0) | -3.7 (4.1)

2. Primary Outcome: Patient Cognitive Test Scores at End of Treatment Period
Description: For cognitive assessment, set of widely used standardized psychometric instruments shown to be sensitive to neurotoxic effects of cancer treatment. Measures assess attention span (Digit Span), graphomotor speed (Digit Symbol), memory (Hopkins Verbal Memory Test-Revised), verbal fluency (Controlled Oral Words Association), visual motor scanning speed (Trail Making Test Part A), executive function (Trail Making Test Part B); motor speed and dexterity (Grooved Pegboard).
Time Frame: Baseline to end of Week 4 treatment period
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years and 11 months
Arm/Group | IR Methylphenidate | SR Methylphenidate | Modafinil
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/10

LIMITATIONS AND CAVEATS:
Early termination lead to limited analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No